CLINICAL TRIAL: NCT03666260
Title: Comparison of the Clinical Effectiveness of the Quadratus Lumborum Block and Femoral Block in the Analgesia of Total Posterior Hip Arthroplasty
Brief Title: Analgesia in Total Hip Arthroplasty by Quadratus Lumborum Block
Acronym: ATHAQLuB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PO18122
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Total Hip Replacement Surgery
Keywords: Total hip replacement surgery; post operative pain; quadratus lumborum block; femoral block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block arm (Experimental)
  Interventions: Procedure: Quadratus Lumborum Block
- Femoral block arm (Active Comparator)
  Interventions: Procedure: femoral block

INTERVENTIONS:
Procedure: Quadratus Lumborum Block — Quadratus Lumborum Block with echography
  Arms: Quadratus Lumborum Block arm
Procedure: femoral block — femoral block with echography
  Arms: Femoral block arm

SUMMARY:
Patients are painful after total hip arthroplasty. These patients have significant co-morbidities. Analgesics cause significant side effects in this population. Locoregional analgesia is therefore an effective means of reducing the consumption of opioids in this surgery.

The "gold standard" of locoregional analgesia after Total Hip Arthroplasty is the femoral block. However, a new technique has recently been described: the Quadratus Lumborum Block.

The comparison of these two techniques is lacking in the literature. The comparison of the Quadratus Lumborum Block to the femoral block in Total Hip arthroplasty is important in the analgesic strategy of patients undergoing this surgery.

DETAILED DESCRIPTION:
The aim of this study is to compare the clinical efficacy of two regional locoregional analgesia strategies in total hip replacement surgery: the ultrasound-guided Quadratus Lumborum Block and the ultrasound-guided femoral block.

This is a double-blind, randomized study in prospective inclusion with a superiority test. Two groups of patients will be compared: a group of patients with a quadratus lumborum block and a group of patients with a femoral block.

Management (quadratus lumborum block or femoral block) will be randomized. The randomization will be stratified on the type of anesthesia (spinal anesthesia and general anesthesia). Randomization will be done on the day of surgery to determine the patient's treatment group. The surgical procedure will not be modified by the participation of the patent in the study.

Patients who would benefit from total hip replacement surgery in the Reims University Hospital and who agreed to participate in the study were included.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for total hip replacement surgery in Reims University Hospital
* Patients agreeing to participate in the research and having signed informed consent
* between 18 yo and 95 yo
* Patients affiliated to a social security system

Exclusion Criteria:

* Patients with allergy to local anesthetics
* Patients with neuropathy
* Patients with an ASA score of 4
* Patients undergoing revision surgery for total hip arthroplasty
* Patients receiving anterior hip total hip replacement surgery
* Patients with a contraindication to the realization of the quadratus lumborum block, femoral block or spinal anesthesia (clinical coagulopathy, infection at the point of puncture ...)
* Patients refusing the proposed techniques

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 24 hours
  Morphine consumption during the 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France